CLINICAL TRIAL: NCT00361608
Title: Monitoring of Nocturnal Hypoglycemia Using EarlySense Monitoring Device
Status: Withdrawn | Type: Observational
Sponsor: EarlySense Ltd. (Industry)
Collaborators: Schneider Children's Medical Center, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: ES-CI 03; 4006
Record Dates: First submitted 2006-08-06; First posted 2006-08-08 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2008-04

CONDITIONS: Type I Diabetes
Keywords: diabetes; hypoglycemia; monitor; children with Type I Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Hypoglycemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Device: EarlySense ES 16

SUMMARY:
This study observes the continuous measurement of breathing patterns, heart rate, restlessness, and tremor in sleep using the EarlySense ES 16 device as a tool in the management of hypoglycemia in pediatric type I diabetes patients.

DETAILED DESCRIPTION:
The study patients are children, 12-18 years old, suffering from type I diabetes. Each patient will participate in the trial for 30 days.

During this period of time the patients' breathing patterns, heart rate, restlessness and tremor in sleep will be measured by the EarlySense device which is put in the patient's bed. These measured values will be compared to:

1. glucose values measured by a "Guardian RT" device - an approved device for CBGM - Continuous Blood Glucose Measurement;
2. glucose levels tested by SBGM -Self Blood Glucose Measurement.

These comparisons will show whether the EarlySense device is applicable in predicting hypoglycemia events in type I diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12-18 years
* Diagnosis of type I diabetes for at least a year
* Home close to participating center
* Guardian able and willing to cooperate with the trial for at least 1 month and prepared to sign the Informed Consent Form.

Exclusion Criteria:

* Recent (within 3 months) admission to emergency room or intensive care unit (ICU) due to any condition unrelated directly to diabetes.
* Any other pre-existing medical pathology unrelated to diabetes.
* Inability of the patient or his guardian to use the Guardian RT.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diabetes I
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liat de Vries, M.D., Principal Investigator — Schneider Children's Medical Center, Israel
Locations (1):
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel